CLINICAL TRIAL: NCT06851208
Title: Do Emotions and Pain Combined Affect Mechanical Pain Thresholds and Other Pain-related Variables in Individuals with Chronic Pain?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Helena Gunnarsson, Dr, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-07781-01 ethic approval
Record Dates: First submitted 2025-02-21; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pain Thresholds; Pain Intensity
Keywords: Pressure pain thresholds; Pain; Emotions
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Within-subjects design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Negative emotion, positive emotion, neutral emotion, control with experimental pain (Experimental): Arm Description: The intervention includes either a negatively emotionally valenced video, a positively emotionally valenced video, a neutrally emotionally valenced video and experimental pain from the cold pressor test that are simultaneosly applied.
  Interventions: Other: Emotional intervention

INTERVENTIONS:
Other: Emotional intervention — Emotional intervention Description: The participant will watch a short video-clip with negative emotional content while simultaneously experience experimentally induced pain.
Other: Emotional intervention — Description: The participant will watch a short video-clip with positive emotional content while simultaneously experience experimentally induced pain.
Other: Emotional intervention — Description: The participant will watch a short video-clip with neutral emotional content while simultaneously experience experimentally induced pain.

SUMMARY:
The purpose of this study is to investigate if different emotional states could influence mechanical pain thresholds and other pain - related variables such as pain tolerance, pain intensity and pain - related negative affect in individuals with chronic pain.

DETAILED DESCRIPTION:
Participants with chronic pain will be randomized into 4 different groups watching different short video-clips (2.20 min), while at the same time experience short-lasting, experimentally induced pain. The negative emotions group will watch an uncomfortable short video containing violence and blood, the positive emotions group will watch a video containing a stand-up comedy show, the neutral emotions group will watch a video about how to paint a house, and the control group will just wait for 2.20 min, without any instructions about what to think about. Pressure pain thresholds, pain tolerance, pain intensity and pain-related negative affect will be measured with an algometer before and after the video-clip combined with experimental pain interventions.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Fluent in Swedish
* Persistent chronic pain with duration > 6 months

Exclusion criteria:

- Known neurological disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pressure pain thresholds | Day 1: baseline PPTs are measured, intervention 2.20 min follows and intervention PPTs are measured directly after the intervention. Recruitment for single appointments for each participant will take place for 4 months.
  Description: Pressure pain thresholds will be measured i kPa with a handheld algometer (Somedic AB).

SECONDARY OUTCOMES:
Pain tolerance (time in seconds the left hand is immersed in cold water 1 degree C). | Day 1: During a single session (30 min), the participant will keep their hand immersed in cold water for as long as possible while watching a video. This time will be measured in seconds.
  Description: The measure pain tolerance equals the time the time the participant keeps their left hand immersed in cold water (1 degree C), before they decide to withdraw their hand. This will be measured in seconds. For each participant, the maximum time to keep the hand immersed in water is 300 seconds. Participants are successively recruited for single appointments for 4 months.
Pain intensity on the NRS | Day 1: Pain intensity will be estimated at single session appointments (30 min) on the NRS (Numerical Rating Scale) after the intervention. Participants will be successively recruited for single session appointments for 4 months.
  Participants will rate their perceived pain intensity on the NRS (Numerical Rating Scale) after the intervention (film-clip combined with pain induction using the cold pressor apparatus with cold water 1 degree C. This will take place on a single session appointment for each participant. Participants will be successively recruited for single session appointments for 4 months.
Pain-related negative affect on the NRS-A | Day 1: Pain intensity will be estimated at single session appointments (30 min) on the NRS-A (Numerical Rating Scale-Anxiety) after the intervention. Participants will be successively recruited for single session appointments for 4 months.
  Description: Perceived pain-related negative affect will be estimated on the NRS-A (Numerical Rating Scale- Anxiety) after the intervention (film-clip combined with pain induction with the cold pressor apparatus with cold water 1 degree C).The pain intensity will be estimated at every single session appointment (30 min) after the intervention on the NRS (Numerical Rating Scale). The participants will be successively recruited for single session appointments for 4 months.

IPD SHARING:
Plan to Share IPD: Undecided